CLINICAL TRIAL: NCT06443567
Title: Arterial Blood Pressure and Cardiac Arrest
Acronym: ABaCAS
Status: Withdrawn | Type: Observational
Why Stopped: Not feasible
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: North West Ambulance Service nhs foundation trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: B01830
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest
Keywords: impedance threshold device; blood pressure; cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- adult cardiac arrest: blood pressure measurement pre and post impedance threshold device placement
  Interventions: Device: impedance threshold device

INTERVENTIONS:
Device: impedance threshold device — impedance threshold device (ResQPOD, Zoll) applied to airway

SUMMARY:
To describe and measure diastolic and systolic femoral arterial pressure during medical cardiac arrest.

To define baseline measures. To describe and measure arterial blood pressure after placement of an ITD device.

To observe the diastolic pressure immediately prior to return of spontaneous circulation.

To quantify and describe the effects of intravenous adrenaline on arterial blood pressure in cardiac arrest.

DETAILED DESCRIPTION:
Cardiac arrest is a complex disorder whose outcome is reliant on a huge number of factors. Moreover, many interventions are time critical, therefore an intervention that may be lifesaving if given early, may have no benefit if instigated further in the disease course. For these reasons' studies involving cardiac arrest are incredibly difficult to carry out and interpret. Many of the interventions carried out during cardiac arrest are aimed at improving blood pressure and thereby increasing the amount of blood and oxygen delivered to the myocardium in the hopes of achieving a return of spontaneous circulation (ROSC). However current data on what a 'normal' blood pressure, based largely upon non-invasive measurement, during cardiac arrest is severely limited, making comparison and evaluation of interventions extremely difficult. This provides the basis for this study in order to prospectively collate and describe data from invasive blood pressure monitoring during adult, medical cardiac arrest in the pre-hospital environment.

3. Research Question/Aim(s) To measure and describe femoral arterial pressure during cardiac arrest with mechanical CPR by a LUCAS device. 3.1 Objectives Primary objective To quantify and describe baseline arterial systolic blood pressure as measured by an invasive femoral line in adult patients suffering medical cardiac arrest in the pre-hospital setting. This will be defined as a line of best fit for systolic blood pressure superimposed on the arterial trace during a 3 minute period.

Secondary Objectives

* To quantify and describe baseline arterial diastolic blood pressure as measured by an invasive femoral line in adult patients suffering medical cardiac arrest in the pre-hospital setting. This will be defined as a line of best fit for diastolic blood pressure superimposed on the arterial trace during a 3 minute period.
* To quantify and describe arterial blood pressure after the placement of an ITD device over a 3 minute period.
* To quantify and describe the effect of intravenous adrenaline on blood pressure as administered in line with ALS guidelines (every 3-5 mins) in adult patients in cardiac arrest.
* To document the diastolic blood pressure of those patients that achieve return of spontaneous circulation (ROSC) following out of hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18years) in medical cardiac arrest
* Deemed suitable to attempt resuscitation.

Exclusion Criteria:

* Prisoners
* <18years
* Pregnancy
* Traumatic cardiac arrest
* Arrest caused by hypovolaemia, tension or tamponade as determined by the clinical team on scene
* Inability to secure a patent airway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18+) suffering an out of hospital cardiac arrest (OHCA) by a presumed medical cause that have been deemed suitable to attempt resuscitation of.
  All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage, and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
systolic femoral invasive blood pressure | 3 mins average with CPR by LUCAS device

SECONDARY OUTCOMES:
femoral diastolic pressure | 3 mins average with CPR by LUCAS device
femoral arterial pressure, both systolic and diastolic | 3 mins average post placement of ICD device

IPD SHARING:
Plan to Share IPD: No